CLINICAL TRIAL: NCT03688126
Title: U.S. Study to Protect Brain Health Through Lifestyle Intervention to Reduce Risk
Acronym: POINTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00052881
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease
Keywords: cognitive decline; dementia; cognitive function
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The U.S. POINTER Coordinating Center (CC) is divided into two distinct entities: the Administrative and Clinical Operations CC and the Data CC. Investigators and staff within the Administrative and Clinical Operations CC will be masked to outcomes data. Investigators and staff within the Data CC will be unmasked to intervention assignment and outcomes. In the clinic, examiners, data entry staff, and the study clinician will be masked to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Guided Lifestyle Intervention (Experimental): Lifestyle modification program that is developed by the participant to meet his/her specific needs.
  Interventions: Behavioral: Self-Guided Lifestyle Intervention
- Structured Lifestyle Intervention (Experimental): Lifestyle modification program that involves participants completing structured activities that target diet, physical exercise, and intellectual and social stimulation.
  Interventions: Behavioral: Structured Lifestyle Intervention

INTERVENTIONS:
Behavioral: Self-Guided Lifestyle Intervention — Lifestyle intervention that involves providing participants with education, support, and tangible tools to assist them in developing and carrying out healthier lifestyle practices.
  Other Names: Self-Guided
  Arms: Self-Guided Lifestyle Intervention
Behavioral: Structured Lifestyle Intervention — Lifestyle intervention that involves a structured program of diet, physical and cognitive exercise, and management of cardiometabolic risks.
  Arms: Structured Lifestyle Intervention

SUMMARY:
The purpose of this research study is to see if lifestyle changes can protect memory and thinking (cognition) as we age. A recent study in Finland found that a combination of physical and cognitive exercise, diet, and social activity protected cognitive function in healthy older adults who were at increased risk of significant memory loss. So far no medications can rival this positive outcome. The point of POINTER is to test if lifestyle change can also protect against memory loss in Americans.

DETAILED DESCRIPTION:
Lifestyle interventions focused on combining healthy diet, physical activity, and social and intellectual challenges may represent a promising therapeutic strategy to protect brain health. The recent results of the population-based 2-year clinical trial, Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER), indicated that a multidomain intervention of physical activity, nutritional guidance, cognitive training, social activities, and management of heart health risk factors protected cognitive function in healthy older adults at increased risk of cognitive decline. As yet, there are no pharmacological treatment options that can rival this effect. Thus, there is an urgent need to expand this work to test the generalizability, adaptability and sustainability of its findings in diverse and global populations. This pivotal U.S. Study to Protect Brain Health through Lifestyle Intervention to Reduce Risk (U.S. POINTER) will test whether a similar 2-year intensive lifestyle intervention, adapted to American culture and delivered within the community, can protect cognitive function in older adults in the U.S. who are at increased risk for cognitive decline and dementia. If successful, the results of this study will have large-scale implications for public policy regarding standard of clinical care and prescriptive practices for a fast-growing and vulnerable population of older adults.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary (not a regular exerciser, determined using the POINTER--modified Telephone Assessment of Physical Activity [TAPA]
* Low MIND Diet score (determined using the MIND Diet Screener)
* No cognitive impairment as per Telephone Interview for Cognitive Status (mTICS) score >32 (includes adjustments for demographics such as age, education and race), the Clinical Dementia Rating Scale (CDR <0.5), and the CDR-Sum of Boxes (CDR-SB <1)
* Risk Score for cognitive decline >2, using the following scoring algorithm:1 point: Suboptimum cardiovascular health (treated or untreated): systolic Blood Pressure >125 mmHg ~OR~ low-density lipoprotein (LDL) cholesterol >115 mg/dL~OR~ glycated hemoglobin (HbA1c) >6.0%1 point: First degree family history (mother, father, sister, brother) of memory impairment- 1 point: Race and ethnicity: African American/Black, Native American, Middle Eastern/North African, or Hispanic/Latinx

  1 point: Older age: 70-79 years 1 point: Sex: male
* Lives in a region where the POINTER interventions will be delivered
* Does not plan to travel outside of the home geographic area for an extended period of time during study participation
* Capacity to complete physical exercise
* Willing to complete all study-related activities for at least 24 months
* Willing to be randomized to either lifestyle intervention group

Exclusion Criteria

* Age <60 or ≥80 years
* Any significant neurologic disease, including any form of dementia, mild cognitive impairment, Parkinson's disease, Huntington's disease, normal pressure hydrocephalus, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma with persistent neurologic sequelae or known structural brain abnormalities
* History of major depression within the last 6 months
* History of bipolar disorder or schizophrenia as per Diagnostic and Statistical Manual (DSM) V criteria
* History of alcohol or substance abuse or dependence within the past 2 years, as per DSM V criteria
* Current or past use of medications for memory impairment or AD (e.g., cholinesterase inhibitors, memantine)
* Current daily use of systemic corticosteroids
* Current use of 3 or more doses of narcotics/week. Use of intermittent narcotics should be stopped 48 hours prior to clinic visits/cognitive testing. Tramadol is allowed as long as the dose remains stable for 3 months.
* Use of psychoactive medications, including benzodiazepines, tricyclic antidepressants, antipsychotics, mood-stabilizers, psychostimulants, anti- parkinsonian medications, anticonvulsant medications or medications with significant central anticholinergic activity are allowed as long as the medication is NOT used to treat an exclusionary medical condition.
* Significant cardiovascular disease (including New York Heart Association (NYHA) Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, or uncontrolled angina)
* Serious conduction disorder (e.g., 3rd degree heart block), uncontrolled arrhythmia, or new Q waves or ST-segment depressions (>3 mm) on ECG (treated atrial fibrillation for more than 1 year or occasional premature ventricular contractions on ECG are not exclusions)
* Myocardial infarction, major heart surgery (i.e., valve replacement, bypass surgery, stent placement, angioplasty), deep vein thrombosis, or pulmonary embolus in the past 6 months
* Large vessel stroke in the past 2 years
* History of transient ischemic attack (TIA) or small vessel stroke in the last 6 months; TIA occurring more than 6 months ago with residual effects
* Current use of insulin to treat type 2 diabetes
* Lung disease requiring either regular use of corticosteroids or the use of supplemental oxygen; intermittent use of corticosteroids or supplemental oxygen to treat chronic obstructive pulmonary disease exacerbation is allowed; use of inhaled steroids for asthma is allowed
* End stage renal disease (e.g., requiring dialysis or as per clinician discretion)
* Clinically significant abnormalities in laboratory blood tests as per judgment of the site Study Clinician
* History within the last 2 years of treatment for primary or recurrent malignant disease, excluding non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with normal prostate-specific antigen post treatment; long-term endocrine therapy for breast cancer is allowed (e.g., tamoxifen, anastrozole)
* History of hip fracture, joint replacement, or spinal surgery in the last 6 months
* Currently receiving physical therapy or cardiopulmonary rehabilitation
* History of a malabsorptive bariatric procedure (gastric bypass, biliopancreatic diversion); other bariatric procedures involving restriction (i.e., sleeve, band) are not exclusionary
* Resides in an assisted living facility or nursing home
* Receives hospice care
* Site PI/Study Clinician discretion regarding medical status, appropriateness of participation or concern about intervention adherence

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Global cognitive function composite score | up to 2 years
  Global cognitive function will be obtained from a composite score derived from subtest scores on the POINTER modified Neuropsychological Test Battery (PmNTB) that includes: Free and Cued Selective Reminding Test, Story Recall, Visual Paired Associates, Number Span, Word Fluency, Trail-Making Test, and Digit Symbol Substitution Test. Scores from each individual test will be converted to z-scores that typically range from -3 to 3, with higher scores reflecting better performance, and averaged to form a composite. The primary outcome is the slope of these composite scores over repeated assessments (standard deviation units per year), with less negative (or positive) slopes reflecting better performance.

SECONDARY OUTCOMES:
Episodic memory composite score | up to 2 years
  This will be a composite score from PmNTB subtests Free and Cued Selective Reminding Test, Story Recall, Visual Paired Associates; and experimental measures: Cogstate One-Card Learning, Face Name Associative Memory Exam, and Behavioral Pattern Separation of Objects, calculated in a manner parallel to how the primary composite outcome is calculated. This secondary outcome is the slope of these composite scores over time (standard deviation units per year) with less negative (or positive) slopes reflecting better performance.
Executive function composite score | up to 2 years
  This will be a composite score from PmNTB subtests Number Span, Word Fluency, Trail-Making Test Part B, Digit Symbol Substitution Test; and experimental measures: Cogstate One Back, and Digital Clock Drawing Test, calculated in a manner parallel to the primary composite outcome is calculated. This secondary outcome is the slope of these composite scores over time (standard deviation units per year) with less negative (or positive) slopes reflecting better performance.
Processing speed composite score | up to 2 years
  This will be a composite score from PmNTB subtests Trail-Making Test Part A and Digit Symbol Substitution Test; and experimental measures: Cogstate Detection and Identification, and Digital Clock Drawing Test calculated in a manner parallel to the primary composite outcome is calculated. This secondary outcome is the slope of these composite scores over time (standard deviation units per year) with less negative (or positive) slopes reflecting better performance.
Clinical dementia rating-sum of boxes | up to 2 years
  The Clinical Dementia Rating (CDR) is a clinical scale that rates the severity of dementia as absent, questionable, mild, moderate, or severe (CDR score of 0, 0.5, 1, 2, or 3, respectively) across six domains. Scores from these domains are summed ranging from 0 to 18, with higher scores reflecting worse performance. The secondary outcome will be the change in the mean scores from baseline to 2 years.
Instrumental activities of daily living (IADL) score | up to 2 years
  The Lawton-Brody IADL is a commonly used scale in clinical practice and research that assess a person's functional ability to complete tasks such as shopping, food preparation, transportation, and managing finances. Scores range from 0 to 8 for women and from 0 to 5 for men, with higher scores reflecting better performance. The secondary outcome will be the change in the mean scores from baseline to 2 years.
Everyday cognition (ECog) score | up to 2 years
  The ECog is a validated scale developed to assess everyday functional status. The short form of the instrument will be used in U.S. POINTER. Scores range from 0 to 4 with higher scores reflecting greater poorer function. The secondary outcome will be the change in the mean scores from baseline to 2 years.
Digital clock drawing test (DCTClock) time | up to 2 years
  DCTClock assesses cognition via novel software that processes information from a commercially available digital pen. This software is able to capture nuances in cognitive performance. Many metrics can be generated with this device. The secondary outcome for U.S. POINTER will be time (in seconds) to completion of the clock drawing test, with longer times reflecting poorer processing speed. The secondary outcome will be the change in the mean scores from baseline to 2 years.
Lifestyle composite score | up to 2 years
  This composite score is based on self-reported Physical Activity Questionnaire, Rush Food Frequency Questionnaire, and the Cognitive Activity Questionnaire. Participants will be ordered with respect to each index, with higher scores reflecting 1) greater daily physical activity, 2) greater conformance with the MIND Diet, and 3) greater cognitive activity. Based on these orderings, participants will be assigned percentiles with respect to each measure relative to the overall group. These percentiles will range from 0 to 100. The secondary outcome will be the average of the three percentiles. The secondary outcome will be the change in the mean scores from baseline to 2 years.
Deficit accumulation frailty index score | up to 2 years
  The Deficit Accumulation Frailty Index (DAFI) is a quantitative measure of frailty that assesses the accumulation of health deficits across various domains, including physical, cognitive, and social functions. The DAFI is calculated by dividing the number of health deficits present by the total number of possible deficits assessed. A score of 0.15 or less is typically considered non-frail, while a score of 0.25 or higher is considered frail. Scores between 0.15 and 0.25 may indicate pre-frailty.

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Baker, PhD, Principal Investigator — Wake Forest University Health Sciences; Mark A Espeland, PhD, Principal Investigator — Wake Forest University Health Sciences; Rachel A Whitmer, PhD, Principal Investigator — University of California, Davis; Miia Kivipelto, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (6):
- United States (6):
  - Northern California, Sacramento, California
  - Chicagoland--Rush, Chicago, Illinois
  - Chicagoland--Advocate Aurora Health, Downers Grove, Illinois
  - North Carolina, Winston-Salem, North Carolina
  - New England--Rhode Island, Providence, Rhode Island
  - Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
The data will be released to national databases upon completion of the study. Links to these databases will be provided at a later time.

REFERENCES:
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Derived] Baker LD, Espeland MA, Whitmer RA, Snyder HM, Leng X, Lovato L, Papp KV, Yu M, Kivipelto M, Alexander AS, Antkowiak S, Cleveland M, Day C, Elbein R, Tomaszewski Farias S, Felton D, Garcia KR, Gitelman DR, Graef S, Howard M, Katula J, Lambert K, Matongo O, McDonald AM, Pavlik V, Raman R, Salloway S, Tangney C, Ventrelle J, Wilmoth S, Willliams BJ, Wing R, Woolard N, Carrillo MC. Structured vs Self-Guided Multidomain Lifestyle Interventions for Global Cognitive Function: The US POINTER Randomized Clinical Trial. JAMA. 2025 Aug 26;334(8):681-691. doi: 10.1001/jama.2025.12923. PMID 40720610
- [Derived] Papp KV, Farias ST, Howard M, Thro A, Ngandu T, Caudle B, Sachs BC, Chan M, Krueger KR, Hartman ERT, Lee A, York MK, Austin MT, Demos KE, Holland TM, Leng X, Raman R, Snyder HM, Carrillo MC, Whitmer RA, Espeland MA, Baker LD; US POINTER Study Group. Baseline cognition and demographic, lifestyle, and cardiovascular risk factors in US POINTER. Alzheimers Dement. 2025 Jul;21(7):e70216. doi: 10.1002/alz.70216. PMID 40667673
- [Derived] Tomaszewski Farias S, Leng I, Papp K, Mehra A, Chan M, York M, Sachs BC, Krueger KR, Lee A, Whitmer R, Snyder HM, Baker LD; U.S. POINTER Study Group. Subjective cognitive decline among diverse older adults: Prevalence and associations with objective cognition. Alzheimers Dement. 2025 Jul;21(7):e70432. doi: 10.1002/alz.70432. PMID 40572055
- [Derived] Espeland MA, Demesie YN, Olson K, Lockhart SN, Farias SET, Cleveland ML, Tangney CC, Crivelli L, Snyder HM, York MK, Baker LD, Whitmer RA, Wing RR, Garcia KR, Callahan KE. Associations Between Deficit Accumulation Frailty and Baseline Markers of Lifestyle in the U.S. POINTER Trial. J Gerontol A Biol Sci Med Sci. 2025 Jan 16;80(2):glae279. doi: 10.1093/gerona/glae279. PMID 39549282
- [Derived] Baker LD, Snyder HM, Espeland MA, Whitmer RA, Kivipelto M, Woolard N, Katula J, Papp KV, Ventrelle J, Graef S, Hill MA, Rushing S, Spell J, Lovato L, Felton D, Williams BJ, Ghadimi Nouran M, Raman R, Ngandu T, Solomon A, Wilmoth S, Cleveland ML, Williamson JD, Lambert KL, Tomaszewski Farias S, Day CE, Tangney CC, Gitelman DR, Matongo O, Reynolds T, Pavlik VN, Yu MM, Alexander AS, Elbein R, McDonald AM, Salloway S, Wing RR, Antkowiak S, Morris MC, Carrillo MC; U.S. POINTER Study Group. Study design and methods: U.S. study to protect brain health through lifestyle intervention to reduce risk (U.S. POINTER). Alzheimers Dement. 2024 Feb;20(2):769-782. doi: 10.1002/alz.13365. Epub 2023 Sep 30. PMID 37776210

DOCUMENTS (1):
  • Informed Consent Form (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03688126/ICF_000.pdf